CLINICAL TRIAL: NCT05811624
Title: Lifestyle Intervention in Overweight/Obese People Suffering From Chronic Low Back Pain: an International Multi-center Randomized Controlled Trial
Brief Title: Lifestyle Intervention in Overweight/Obese Chronic Low Back Pain (CLBP) Patients: an International Multi-center RCT
Acronym: BO2WL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Bern University of Applied Sciences (Other); University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Jo Nijs, Full professor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BUN1432022000296; G094322N (Other Grant/Funding Number: Research Foundation Flanders); 2022-02210 (Other: Ethical Committee Switzerland (Bern)); S011866-42-PHYW (Other Grant/Funding Number: Swiss National Science Foundation (SNSF))
Record Dates: First submitted 2023-03-14; First posted 2023-04-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Overweight or Obesity; Chronic Low-back Pain
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized (1/1) into one of the two treatment arms (control or intervention)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Intervention (Experimental): Physiotherapy intervention, including behavioral weight reduction program combined with pain neuroscience education and cognition-targeted exercise therapy.
  Interventions: Behavioral: Physiotherapy intervention, including behavioral weight reduction program combined with pain neuroscience education and cognition-targeted exercise therapy.
- Control Intervention (Active Comparator): Physiotherapy intervention, including pain neuroscience education and cognition-targeted exercise therapy alone.
  Interventions: Behavioral: Physiotherapy intervention, including pain neuroscience education and cognition-targeted exercise therapy alone.

INTERVENTIONS:
Behavioral: Physiotherapy intervention, including behavioral weight reduction program combined with pain neuroscience education and cognition-targeted exercise therapy. — 14 weeks, 18 treatment sessions
  This includes:
  * 3 sessions of Pain Neuroscience Education during the first two weeks (of which the second one will be held online). The aim is to to reconceptualize pain, to increase pain coping skills and to convince the patients that pain is in the brain, and that hypersensitivity of the central nervous system rather than local tissue damage contributes to their symptoms.
  * 15 sessions which will focus simultaneously on cognition-targeted exercise therapy and behavioral weight reduction. The aim of the exercise program is to confront the patient with movements and activities that are feared, avoided and/or painful. The behavioral weight reduction program includes a lifestyle approach, with changes in diet, behavior, and a physical exercise weight loss program, all aiming for a caloric deficit of 500 to 700 kcal/day.
  Other Names: EXP (Experimental intervention)
  Arms: Experimental Intervention
Behavioral: Physiotherapy intervention, including pain neuroscience education and cognition-targeted exercise therapy alone. — 14 weeks, 18 treatment sessions
  This includes:
  * 3 sessions of Pain Neuroscience Education during the first two weeks (of which the second one will be held online). The aim is to to reconceptualize pain, to increase pain coping skills and to convince the patients that pain is in the brain, and that hypersensitivity of the central nervous system rather than local tissue damage contributes to their symptoms.
  * 15 sessions which will only focus on cognition-targeted exercise therapy. The aim of the exercise program is to confront the patient with movements and activities that are feared, avoided and/or painful.
  Other Names: CON (Control intervention)
  Arms: Control Intervention

SUMMARY:
Chronic low back pain (CLBP) is the most expensive cause of workrelated disability: it causes the highest number of years lived with disability. The most severe and debilitated CLBP patients often have comorbidities such as overweight and obesity. Despite the growing body of scientific literature pointing towards the close interaction between overweight/obesity and CLBP, few treatment programs for people with CLBP nowadays take overweight into account. Therefore this study will examine the added value of a behavioral weight reduction program (changes in diet, behavior and physical exercise) to current best evidence rehabilitation (pain neuroscience education plus cognition-targeted exercise therapy) for overweight or obese people with CLBP. An international, multicenter randomized controlled trial comparing a behavioral weight reduction program combined with pain neuroscience education and cognition-targeted exercise therapy versus pain neuroscience education and cognition-targeted exercise therapy alone, will be conducted. The primary outcome is pain and the primary endpoint was chosen at 12 months follow-up; secondary outcomes include health care use and daily functioning (see detailed description of outcomes for an overview of all secondary outcomes). If the promising results of the proof of concept study are corroborated, the new intervention will have a high socio-economic impact, including an annual health care cost reduction of €66 million in Switzerland, and €60 million in Flanders, and is expected to increase life expectancy in the long term.

DETAILED DESCRIPTION:
Rationale:

Chronic low back pain (CLBP) is the most common and important clinical, social, economic, and public health problem of all chronic pain disorders across the world. In addition to its high prevalence, CLBP is a severely disabling disorder characterized by tremendous personal and socioeconomic impact. Furthermore, it is the most common cause of work-related disability, generating long-term sick-leaves, and it causes the highest number of years lived with disability.

The most severe and debilitated CLBP patients often have comorbidities such as overweight and obesity. In fact, pain intensity and disability in people with CLBP show dose-responses to body mass index (BMI), waist circumference, percent fat and fat mass. Ample studies and several meta-analyses indeed confirm that overweight and obesity are associated with LBP, with overweight and obesity even being a risk factors for low back pain. Regarding socio-economic impact, overweight or obesity is not only related to LBP persistence, but also to higher rates of health care seeking for LBP. Obviously, people with CLBP who are overweight or obese, are likely to have more complex health needs requiring focus on lifestyle behavioral factors such as physical activity/exercise and diet.

CLBP is a complex disorder which is difficult to treat. Exercise therapy is an evidence-based treatment for CLBP both general exercises and cognition-targeted exercise therapy have shown beneficial effects on pain in patients with CLBP. Unfortunately, current treatments for CLBP apply a 'one-size-fits-all' approach and do not address comorbidities like obesity. This knowledge gap is now acknowledged internationally: overweight and obesity are increasingly recognized as a plausible therapeutic target for people with CLBP. Despite the growing body of scientific literature pointing towards the close interaction between overweight/obesity and CLBP few treatment programs for people with CLBP nowadays take overweight into account.

Few studies explored the added value of weight reduction to the management of people with CLBP. Yet, proof of concept for combining dietary changes with exercise therapy for patients with CLBP and comorbid overweight/obesity show promising results. Here we propose studying the added value of a behavioral weight reduction program (changes in diet, behavior, and physical exercise) to blended rehabilitation (PNE plus CTET) for overweight or obese people with CLBP. Both treatments are effective in their specific target population (i.e., behavioral weight reduction for overweight/obese people and PNE plus CTET for people with CLBP and normal BMI), but whether their combined approach is cumulative in overweight/obese people with CLBP is currently unknown and represents an important research priority.

Objectives:

The primary objective is to examine if a behavioral weight reduction program combined with Pain Neuroscience Education (PNE) and Cognition-Targeted Exercise Therapy (CTET) is superior to reduce pain at 12 months follow-up compared PNE and CTET alone, in overweight or obese people with CLBP.

Secondary objectives are to examine the effects of adding a behavioral weight reduction program combined with PNE and CTET, compared to PNE and CTET alone, on 1) other pain related outcomes (pain interference, pain distribution and pain beliefs), 2) on anthropometrics (body weight/composition, muscle thickness and fat distribution), 3) on energy balance related behavior (24h continuous activity monitoring, dietary intake and sleep) and finally 4) on health economics (heath care utilization, productivity loss and quality of life) at 12 months follow-up.

Interventions:

Both interventions (experimental and control) are organized equally: all participants will receive 18 treatment sessions over a 14-week period see table 2 for a detailed overview. Rather than practical, treatment arms will differ in content.

The control intervention will consist of a total of 18 treatment sessions distributed over 14 weeks. It comprises of only the chronic-pain-focused interventions: 3 sessions of PNE in the first 2 weeks & secondly, 15 sessions of CTET in the remaining 12 weeks.

The experimental intervention will consist of a total of 18 treatment sessions distributed over 14 weeks. The first part will consist of chronic-pain-focused interventions: firstly, 3 sessions of PNE in the first 2 weeks & secondly, 15 sessions of CTET in the remaining 12 weeks. The second part will consist of a more weight-reduction-focused intervention. The weight reduction intervention is a lifestyle approach that will be integrated in the CTET intervention, implying that grading daily physical activity and exercise levels will aim at reducing weight (i.e. together with a change in diet we aim at a caloric deficit of 500 to 700 kcal/day) and improving pain cognitions at the same time.

Study design:

Randomized controlled trial with follow-up assessments directly post-treatment (T1), 3 months post-treatment (T2), 6 months post-treatment (T3), 9 months post-treatment (T4) and 12 months post-treatment (T5).

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 - 65 years)
* Overweight (BMI ≥ 25 kg/m2) or obese (BMI ≥ 30 kg/m2) women and men.
* CLBP (n=252), which is defined as nonspecific low back pain for at least 3 months duration, currently seeking care for low back pain and leg pain not ≥ 7 (on a maximum of 10) on a numeric rating scale.
* Continue usual care 6 weeks prior to (to obtain a steady stat) and during study participation.
* Depending on the country of inclusion: Native Dutch speaker (for Belgium) or Native German speaker (for Switzerland).

Exclusion Criteria:

* Patients with BMI ≥ 40 kg/m² will be excluded as people being morbid obese are eligible to undergo abdominal surgery. Because BMI may not always correspond to the same body fat percentage in different individuals (e.g., athletic types with higher muscle mass may also have BMIs ≥ 25 km/kg²), each participant's body fat percentage will be measured using the TANITA and compared to the body fat percentage reference values. Participants with exceeding BMI but falling into the healthy fat percentage range (which is sex-, age- and ethnicity dependent will be excluded.
* Pregnant, currently breastfeeding or given birth in preceding year.
* Currently receiving dietary or exercise interventions or received in the past 6 weeks.
* Show evidence of specific spinal pathology based on self-report (e.g., hernia, spi-nal stenosis, spondylolisthesis, infection, spinal fracture or malignancy), or a se-vere underlying comorbidity specific diagnoses that interfere with treatment (e.g., diagnosed diabetes, cardiovascular problems, metabolic diseases)
* Other severe diseases based on current medication intake or being currently treated by a medical doctor for a specific diagnosis, (e.g. diagnosed eating disorders).
* Ongoing problems or cases with insurance companies regarding their back.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory - Average pain Intensity | Change from baseline to 12 months post-intervention
  Since CLBP is a fluctuating condition, the question "please rate your pain by circling the one number that best describes your pain on the AVERAGE" is used as primary outcome measure to evaluate pain intensity. The answer to this question is formulated on an 11-point (i.e., 0-10, a decrease of 30% is considered as clinically significant) numeric rating scale (NRS). Higher scores indicate higher pain intensity.

SECONDARY OUTCOMES:
Brief Pain Inventory - Pain intensity (Average, worst, least, now) | This outcome will be assessed at Baseline, directly post-treatment, 3 months post-treatment, 6 months post-treatment and 12 months past-treatment
  The BPI will also be used to assess pain intensity at other timepoints.
Brief Pain Inventory - Pain interference on functioning | This outcome will be assessed at Baseline, directly post-treatment, 3 months post-treatment, 6 months post-treatment and 12 months past-treatment
  The BPI also evaluates the impact of pain on functioning. The BPI measures how much pain interferes with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep on an 11-point NRS (ranging from 0-10). Higher scores indicate a bigger interference of pain with activities of daily life.
Pain distribution and pain extent by pain drawings | This outcome will be assessed at Baseline, directly post-treatment, and 12 months past-treatment
  Extent of pain will be indicated by the participants making use of a digital pain drawing obtained using a digital tablet and commercially available sketching software
Tampa Scale for Kinesiophobia (TSK) | This outcome will be assessed at Baseline, directly post-treatment, 3 months post-treatment, 6 months post-treatment and 12 months past-treatment
  The TSK contains questions about pain-related fear of movement, fear of (re)injury and fear avoidance behavior. The TSK results in a score ranging from 17 to 68, where higher scores indicate an increasing degree of kinesiophobia.
Fear Avoidance Belief Questionnaire | This outcome will be assessed at Baseline, directly post-treatment, 3 months post-treatment, 6 months post-treatment and 12 months past-treatment
  The fear avoidance belief questionnaire focuses on LBP patient's beliefs about how physical activity and work affect LBP (fear of pain caused by physical activity). This questionnaire results in a total score (ranging from 0 to 96) and two subscale scores: work subscale (ranges from 0 to 42) and physical activity subscale (score 0 to 24). Higher scores indicate more strongly held fear avoidance beliefs.
Body weight - Tanita | This outcome will be assessed at Baseline, directly post-treatment, and 12 months past-treatment
  Body weight (kg) will be measured using TANITA MC-780SMA Bio-electrical Impedance Analyzer.
BMI - Tanita | This outcome will be assessed at Baseline, directly post-treatment, and 12 months past-treatment
  BMI will be measured using TANITA MC-780SMA Bio-electrical Impedance Analyzer.
Fat mass - Tanita | This outcome will be assessed at Baseline, directly post-treatment, and 12 months past-treatment
  Fat mass will be measured using TANITA MC-780SMA Bio-electrical Impedance Analyzer.
Fat free mass - Tanita | This outcome will be assessed at Baseline, directly post-treatment, and 12 months past-treatment
  Fat free mass will be measured using TANITA MC-780SMA Bio-electrical Impedance Analyzer.
Muscle mass - Tanita | This outcome will be assessed at Baseline, directly post-treatment, and 12 months past-treatment
  Muscle mass will be measured using TANITA MC-780SMA Bio-electrical Impedance Analyzer.
Body Water - Tanita | This outcome will be assessed at Baseline, directly post-treatment, and 12 months past-treatment
  Body water will be measured using TANITA MC-780SMA Bio-electrical Impedance Analyzer.
Waist-hip circumference | This outcome will be assessed at Baseline, directly post-treatment, and 12 months past-treatment
  Measured using a Cescorf measuring tape,
Regional body composition - portable ultrasound scanner | This outcome will be assessed at Baseline, directly post-treatment, and 12 months past-treatment
  Subcutaneous adipose tissue thickness of the triceps, biceps, subscapular, iliac crest, supraspinal, abdominal and medial calf will be assessed. Additionally, muscle thickness of the multifidi will be assessed.
Accelerometry Fitbit | This outcome will be assessed at Baseline, directly post-treatment, and 12 months past-treatment
  To objectively measure sedentary behavior, physical activity and sleep quantity/quality
Sleep Quality - Pittsburg Sleep Quality Index | This outcome will be assessed at Baseline, directly post-treatment, 3 months post-treatment, 6 months post-treatment and 12 months past-treatment
  Questionnaire assessing Sleep Quality. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Dietary Intake | This outcome will be assessed at Baseline, directly post-treatment, 3 months post-treatment, 6 months post-treatment and 12 months past-treatment
  a 3 day food diary, 2 week days and 1 weekend day, will be used to analyse their dietary intake.
Health Economics - Medical Consumption Questionnaire | This outcome will be assessed at Baseline, directly post-treatment, 3 months post-treatment, 6 months post-treatment, 9 months post-treatment and 12 months past-treatment
  a generic instrument for measuring patient's total direct and indirect medical consumption. For this type of questionnaire and the aspect it is measuring, we cannot refer to minimum or maximum values.
Health Economics - Productivity Cost Questionnaire | This outcome will be assessed at Baseline, directly post-treatment, 3 months post-treatment, 6 months post-treatment, 9 months post-treatment and 12 months past-treatment
  to obtain data regarding the indirect medical costs (e.g., the costs due to absenteeism or presenteeism). For this type of questionnaire and the aspect it is measuring, we cannot refer to minimum or maximum values.
Health Economics - EuroQol EQ-5D-5L | This outcome will be assessed at Baseline, directly post-treatment, 3 months post-treatment, 6 months post-treatment, 9 months post-treatment and 12 months past-treatment
  to assess health profiles which will be transformed into utilities using the Flemish or German Tariffs respectively. For this type of questionnaire and the aspect it is measuring, we cannot refer to minimum or maximum values.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (2):
- Vrije Universiteit Brussel, Brussels, Belgium
- Berner Fachhochschule, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
We do not plan to share any IPD

REFERENCES:
- [Derived] Schurz AP, Lutz N, Liechti M, Malfliet A, Vanroose M, Maebe Z, Nijs J, Van Bogaert W, Clarys P, Clijsen R, Baur H, Taeymans J, Deliens T. Cost of illness analysis in individuals with overweight or obesity and chronic low back pain in the Bern metropolitan area (the BO2WL trial). Front Public Health. 2026 Jan 13;13:1705891. doi: 10.3389/fpubh.2025.1705891. eCollection 2025. PMID 41607914
- [Derived] Schurz AP, Deliens T, Liechti M, Vanroose M, Clijsen R, Nijs J, Malfliet A, Van Bogaert W, Clarys P, Baur H, Taeymans J, Lutz N. Economic evaluation of a lifestyle intervention for individuals with overweight or obesity suffering from chronic low back pain (the BO2WL trial): a protocol for a health economic analysis. BMJ Open. 2025 Jun 20;15(6):e098272. doi: 10.1136/bmjopen-2024-098272. PMID 40541436